CLINICAL TRIAL: NCT03374982
Title: Effect of the DentalVibe Injections System on Pain During Local Anesthesia Injections in Children
Brief Title: Effect of the DentalVibe Injection System on Pain During Local Anesthesia Injections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0661-17-FB
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized cross-over clinical trial wherein the study subject serves as his or her own control.
Who Masked: Outcomes Assessor
Masking Description: The person administering the FACES pain rating scale will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DentalVibe turned On then turned Off (Experimental): DentalVibe will be turned on during local anesthetic injection at the first appointment. DentalVibe will be turned off during local anesthetic injection at the second appointment.
  Interventions: Device: DentalVibe
- DentalVibe turned Off and then turned On (Experimental): DentalVibe will be turned off during local anesthetic injection at the first appointment. DentalVibe will be turned on during local anesthetic injection at the second appointment.
  Interventions: Device: DentalVibe

INTERVENTIONS:
Device: DentalVibe — The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.

SUMMARY:
Title: Effect of the DentalVibe injection system on pain during local anesthesia injections in children.

Purpose: The purpose of this study is to compare self-reported pain scale measurements using the Wong-Baker FACES pain rating scale from an experimental group (local anesthesia injection with DentalVibe system) and a control group (traditional local anesthesia injection with DentalVibe system turned off) in children.

Eligibility: Children age 5-11 years old who require local anesthesia for bilateral dental treatment at University of Nebraska Medical Center (UNMC) pediatric dental clinic. Children must understand and speak English.

Interventions and evaluations: Each patient will have two separate restorative appointments where the DentalVibe will be used during local anesthetic injections. One appointment the DentalVibe will be turned on and one appointment the DentalVibe will be turned off. After each injection the child will be shown the Wong Baker FACES Pain Rating Scale and asked to pick a face associated with their level of hurt during the injection.

Follow-up: All children will be followed up with any necessary recommended dental treatment.

DETAILED DESCRIPTION:
Up to 50 children between the ages of 5-11 years will participate in this randomized, controlled, cross-over, split-mouth study. There will be no gender restrictions used in this study. Participants will be recruited from a continuous sample of patient seen at the UNMC pediatric dental clinic and will be selected based on their need for dental treatment. Each child will have 2 separate dental appointments.

Written consent will be obtained from parent or guardian prior to first restorative appointment. Verbal consent will be obtained prior to second restorative appointment.

Dr. Marshall will be the provider for every patient. The same dental assistant will be used for each appointment. All treatment will be completed in the same private quiet room. Both Dr. Marshall and the dental assistant will wear the same color scrubs and black lab jackets during all appointments.

One appointment patient will receive local anesthetic dental injection with the DentalVibe turned on and at one appointment the child will receive local anesthetic dental injection with the DentalVibe off. Used strictly as a check/lip retractor. The child will be randomly assigned via a random number generator to either the DentalVibe on or off during the initial appointment. During the DentalVibe turned on appointment, the DentalVibe will be introduced to each child to make him/her familiar with the vibration sensation.

All patients will receive 5 mins of O2, then nitrous oxide (N2O) will be titrated up to 50%N2O/50%O2. When appointment is complete the child will receive 5 mins of 100% O2.

At both restorative appointment a cotton tip applicator with 20% Benzocaine topical anesthetic gel (Patterson) will be administered for 1 min. 2% Lidocaine hydrochloride (HCl) with 1:100,000epinepherine (Patterson Dental) will the be deposited using a medium-length (0.4mm) with 27-gauge short needles. Local anesthetic injections will be referred to as "sleepy juice." Buccal and lingual infiltration will perform on the maxilla. Mandibular blocks will be performed on the mandible. One cartridge of local anesthetic will be used at each appointment. After administration, patient will be shown the Wong Baker FACES pain rating scale and asked to rate the amount of discomfort experienced during the injection by pointing to the face or number. The following manuscript will be used:

"Each face represents a person who has no hurt, or some hurt, or a lot of hurt." "Face 0 doesn't hurt at all. Face 2 hurts just a little bit. Face 4 hurts a little bit more. Face 6 hurts even more. Face 8 hurts a whole lot. Face 10 hurts as much as you can imagine, although you don't have to be crying to have this worst pain." "Touch the face of the hurt you felt when I gave you the sleepy juice."

After child has rated pain Dr. Marshall will continue with restorative treatment. The same process will be followed at the second appointment. Appointments will be scheduled 3-4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 5-11 who require dental treatment that requires bilateral local anesthesia on the maxilla or mandible. Subjects must understand and speak English.

Exclusion Criteria:

* No children with presence of medically or developmentally compromising conditions (autism, cerebral palsy, moderate/severe asthma); history of chronic disease (seizure disorder, cardiac disorder, hematological disease, endocrine disorder, liver disease, renal disease). Non-English speakers will be excluded. Subject who require oral sedation or general anesthesia for treatment due to behavior or medical history will be excluded.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Johnson, DDS, Principal Investigator — University of Nebraska
Locations (1):
- Children's Hospital & Medical Center Specialty Pediatric Center Dental Clinic, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DentalVibe Turned On and Then Turned Off: DentalVibe will be turned on during local anesthetic injection at the first appointment. DentalVibe will be turned off at the second appointment
  DentalVibe: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
- DentalVibe Turned Off and Then Turned On: DentalVibe will be turned off during local anesthetic injection at the first appointment. DentalVibe will be turned on at the second appointment
  DentalVibe: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
Period: Overall Study
Arm/Group | DentalVibe Turned On and Then Turned Off | DentalVibe Turned Off and Then Turned On
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DentalVibe On, Then Off: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
  DentalVibe will be turned on during local anesthetic injection at first assigned appointment, then off at second appointment.
- DentalVibe Off, Then On: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
  DentalVibe will be turned off during local anesthetic injection at first assigned appointment, then on at second appointment.
- Total: Total of all reporting groups
Arm/Group | DentalVibe On, Then Off | DentalVibe Off, Then On | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Customized [Count of Participants; unit: Participants]
  Age (5-11 years) | 12 | 11 | 23
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/gender not recorded Population: Sex/gender not recorded
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Pain Rating Using Wong-Baker FACES Scale
Description: The scale includes pictures of facial expressions with correlating numerical scale of 0-10. 0 being no hurt and 10 being the worst hurt.
Time Frame: Immediately after local anesthetic delivery
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DentalVibe On: DentalVibe will be turned on during local anesthetic injection at one appointment.
  DentalVibe: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
- DentalVibe Off: DentalVibe will be be turned off during local anesthetic injection at one appointment.
Arm/Group | DentalVibe On | DentalVibe Off
Number analyzed (Participants) | 23 | 23
score on a scale | 3.57 (3.13) | 5.13 (3.40)

ADVERSE EVENTS:
Time Frame: During procedure, up to 1 hour at each visit (2 visits)
Groups:
- DentalVibe On: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
  DentalVibe will be turned on during local anesthetic injection at first or second randomly assigned appointment.
- DentalVibe Off: The DentalVibe is a handheld device that delivers vibration to the tissue during local anesthetic administration.
  DentalVibe will be turned off during local anesthetic injection at the other appointment (based on randomization).
Arm/Group | DentalVibe On | DentalVibe Off
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03374982/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03374982/ICF_001.pdf